CLINICAL TRIAL: NCT02154100
Title: Tart Cherry Improves Cardiovascular Risk Factors Associated With Metabolic Syndrome
Brief Title: Tart Cherry, Metabolic Syndrome, and Cardiovascular Risk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Cherry Research Committee (Other)
Responsible Party: Principal Investigator, Bahram Arjmandi, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF02406
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Metabolic Syndrome; Cardiovascular Diseases; Diabetes
Keywords: Metabolic Syndrome; Arterial Stiffness; Blood Pressure; Endothelial Function; Tart Cherries
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tart Cherry (Experimental): 12 weeks of tart cherry juice taken in two doses of 240 ml per day.
  Interventions: Dietary Supplement: Tart Cherry
- Placebo (Placebo Comparator): 12 weeks tart cherry juice taken in two doses of 240 ml per day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Tart Cherry — 12 weeks of tart cherry juice taken in two doses of 240 ml per day.
  Arms: Tart Cherry
Dietary Supplement: Placebo — 12 weeks of tart cherry juice taken in two doses of 240 ml per day.
  Arms: Placebo

SUMMARY:
The hypothesis of this study is that the daily consumption of 480 ml tart cherry juice for twelve weeks will improve blood pressure and arterial stiffness by improving endothelial-mediated vasodilation and vascular sympathetic activity and favorably altering biochemical markers associated with cardiovascular risk. 28 men and women between the ages of 20 and 40 who have three of the five features of metabolic syndrome as defined by the Adult Treatment Panel III will be included in the study. After a two-week run-in phase, eligible men and women will be randomly assigned to one of two treatment groups: 1) 480 ml tart cherry juice or 2) 480 ml control drink daily for twelve weeks. After an initial telephone screening, all participants will be requested to report to the study site for their first visit. On the first visit (screening), participants will be provided with verbal and written explanation of the project. They will then be asked to sign an informed consent form, followed by measuring waist circumference, resting brachial blood pressure, fasting serum triglycerides, high density lipoprotein cholesterol, and glucose levels to confirm metabolic syndrome. Baseline assessments will be performed for medical history, medication use, dietary intake, and physical activity. Qualified participants will be scheduled for their second visit two weeks later (actual baseline data collection) and randomly assigned to their treatment group. On the second (baseline) visit between the hours of 7-10 A.M., blood pressure and vascular function will be measured followed by blood draw. Anthropometrics will be measured. Participants will be provided with their assigned treatment and will receive standard instructions on how to fill out daily diaries for their treatment, and for food and physical activity records. Blood pressure, vascular function, blood draw, and anthropometric, body composition, diet, and physical activity assessments will be repeated at 6- (third visit), and 12-week (final visit) intervals. All cardiovascular measurements will be performed between 7:00 to 10:00 A.M., in a quiet temperature-controlled room in the supine position after an overnight fast and 12 hours after the abstinence of caffeine and/or 24 hours after the last bout of moderate to heavy physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Three of the following five features at the screening visit:
* Waist circumference of ≥ 40 inches for men and 35 inches for women
* Serum triglycerides ≥ 150 mg/dL
* Serum high density lipoprotein cholesterol levels < 40 mg/dL for men and <50 mg/dL for women
* Blood pressure ≥ 130/85 mm Hg
* Fasting blood glucose level ≥ 110 mg/dL

Exclusion Criteria:

* Taking hypoglycemic, antihypertensive or cholesterol-lowering medications
* Diagnosed cardiovascular disease
* Uncontrolled hypertension (≥ 160/100 mmHg)
* Diabetes mellitus
* Other active chronic diseases such as cancer, asthma, glaucoma, thyroid, kidney, liver and pancreatic disease
* Participating in a weight loss program
* Heavy smokers (> 20 cigarettes per day)
* Heavy drinkers (> 12 alcoholic drinks per week)
* Abnormal menstrual cycle

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 12 weeks
  By measuring brachial and aortic blood pressure at rest and during physiological stress (handgrip exercise and post-exercise muscle ischemia).
Arterial Stiffness | 12 weeks
  By measuring arterial stiffness and augmentation index at rest and during physiological stress (handgrip exercise and post-exercise muscle ischemia).

SECONDARY OUTCOMES:
Autonomic Control of Blood Pressure | 12 weeks
  By measuring blood pressure variability and baroreflex sensitivity at rest and during physiological stress.
Endothelial Function | 12 weeks
  By measuring markers of endothelial function.
Endothelial-mediated Vasodilation | 12 weeks
  By measuring flow-mediated dilation in the brachial artery.
Inflammation | 12 weeks
  By measuring a marker of inflammation.
Oxidative Stress | 12 weeks
  By measuring markers of oxidative stress.
Insulin Sensitivity | 12 weeks
  By measuring fasting glucose, insulin, and homeostatic model assessments of insulin resistance, sensitivity, and beta cell function.
Atherogenic Markers | 12 weeks
  By measuring adhesion factors, lipid profiles, and atherogenic risk ratios.
Body Composition | 12 weeks
  By measuring fat mass and fat-free mass using dual-energy X-ray absorptiometry and anthropometrics.

CONTACTS AND LOCATIONS:
Overall Officials: Bahram H. Arjmandi, PhD, RD, Principal Investigator — Department of Nutrition, Food and Exercise Sciences, Center for Advancing Exercise and Nutrition Research on Aging, Florida State University; Arturo Figueroa, MD, PhD, Principal Investigator — Department of Nutrition, Food and Exercise Sciences, Florida State University; Sarah A. Johnson, PhD, RDN, Principal Investigator — Department of Food Science and Human Nutrition, Colorado State University
Locations (1):
- Department of Nutrition, Food and Exercise Sciences, Center for Advancing Exercise and Nutrition Research on Aging, Florida State University, Tallahassee, Florida, United States